CLINICAL TRIAL: NCT06989801
Title: Benefits of a Nature Walk vs. an Urban Walk in Reducing Depressive Symptoms: A Randomized Controlled Study Among College Students
Brief Title: Benefits of Outdoor Walks in Reducing Depressive Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Xuanyi Wang, PhD Student, Department of Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00022242
Record Dates: First submitted 2025-04-11; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants were informed that the study was about outdoor walking interventions but were not told about the different groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Urban Walk (Active Comparator): Regular walks in an urban area, 30 minutes twice a week for 3 weeks.
  Interventions: Behavioral: Urban Walk
- Nature Walk (Experimental): Regular walks in a natural area, 30 minutes twice a week for 3 weeks.
  Interventions: Behavioral: Nature Walk
- Active Nature Walk (Experimental): Regular walks in a natural area, 30 minutes twice a week for 3 weeks. Prior to the walk, participants will be instructed to actively interact with the natural environment.
  Interventions: Behavioral: Active Nature Walk

INTERVENTIONS:
Behavioral: Urban Walk — For each session, participants will take a 30-minute walk in an urban environment along a designated looped route. They will walk at a comfortable pace and follow the assigned path. During the walk, participants will be instructed to experience their surroundings as naturally as possible. No specific activities beyond walking are required.
  To fully immerse in the experience, participants will be asked to avoid using their phones unless necessary (e.g., in case of an emergency). They should keep the GPS app recording throughout the walk without interacting with it-just allow it to run in the background.
  Once the loop is completed, participants will stop the GPS recording and return to the starting point, where a research team member will be waiting. They will then be guided indoors to complete a brief post-walk survey and participate in a short interview to share their experience.
  Arms: Urban Walk
Behavioral: Nature Walk — For each session, participants will take a 30-minute walk in a natural environment along a designated looped route. They will walk at a comfortable pace and follow the assigned path. During the walk, participants will be instructed to experience their surroundings as naturally as possible. No specific activities beyond walking are required.
  To fully immerse in the experience, participants will be asked to avoid using their phones unless necessary (e.g., in case of an emergency). They should keep the Gaia GPS app recording throughout the walk without interacting with it-just allow it to run in the background.
  Once the loop is completed, participants will stop the GPS recording and return to the starting point, where a research team member will be waiting. They will then be guided indoors to complete a brief post-walk survey and participate in a short interview to share their experience.
  Arms: Nature Walk
Behavioral: Active Nature Walk — For each session, participants will take a 30-minute walk in a natural area, following a designated looped route. Unlike a regular walk, participants will be encouraged to engage with nature (e.g., listening to natural sounds, looking for birds, and touching flowers).
  To make the most of the walk, participants will be asked to avoid using their phones unless necessary (e.g., in case of an emergency). They should keep the Gaia GPS app recording throughout the walk without interacting with it-just letting it run in the background.
  Once the loop is completed, participants will stop the GPS recording and return to the starting point, where a research team member will be waiting. They will then be guided indoors to complete a brief post-walk survey and participate in a short interview to share their experience.
  Arms: Active Nature Walk

SUMMARY:
The goal of this clinical trial is to determine whether outdoor walking in different environments-urban or natural-can reduce depressive symptoms among college students. The study also tests whether providing prompts for active engagement during nature walks enhances the benefits compared to unstructured nature walks.

Participants will be randomly assigned to one of three groups: (1) urban walk, (2) nature walk, or (3) active nature walk with guided interaction. Each participant will walk for 30 minutes, twice a week, for 3 weeks, complete questionnaires, and participate in interviews.

Our primary outcome (PHQ-9) will be used to test the following two primary hypotheses:

* Hypothesis 1: Participants in both nature walk conditions (combined) will show greater reductions in depressive symptoms (PHQ-9) than those in the urban walk group.
* Hypothesis 2: Participants in the active nature walk will show greater reductions than those in the regular nature walk.

DETAILED DESCRIPTION:
The investigators aim to compare how walking in different outdoor environments influences depressive symptoms among college students. Specifically, the investigators will assess:

1. walking in an urban environment (like a busy city street),
2. walking in a natural environment regularly (e.g., walking without specific guidance), and
3. walking in a natural environment with guided interaction prompts (e.g., noticing birds, listening to sounds, touching flowers).

Standardized questionnaires will measure changes in depressive symptoms, anxiety, affect, cognitive flexibility, nature connection, and Presence across all three groups.

The investigators will also explore potential mechanisms behind any observed effects, including interaction patterns, presence, cognitive changes, and emotional responses to the different environments.

ELIGIBILITY:
Inclusion Criteria:

* College students in Seattle
* Aged over 18.
* Having depressive symptoms with self-rated Patient Health Questionnaire-9 (PHQ-9) scored higher than 5.
* Normal or corrected-to-normal visual acuity.
* No identified hearing impairment.
* No history of neurological or mental disorders.

Exclusion Criteria:

* Receiving clinical psychiatric treatment or psychological counseling.
* Failing in providing consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-12-17 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire | Right before the first walking session, immediately after the sixth walking session, and one month after the sixth walking session.
  Patient Health Questionnaire measures the severity of depressive symptoms. It includes nine items that evaluate symptoms such as persistent sad, loss of interest or pleasure in activities, fatigue, and lack of energy. Each item is rated on a 4-point Likert scale, ranging from 0 (not at all) to 3 (nearly every day). Higher scores indicate more severe symptoms of depression.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 7-item scale | Right before the first walking session, immediately after the sixth walking session, and one month after the sixth walking session.
  Generalized Anxiety Disorder 7-item scale measures the severity of anxiety. It includes seven items, such as persistent nervousness, excessive worrying, difficulty relaxing, feeling restless, and becoming easily irritated. Each item is rated on a 4-point Likert scale, ranging from 0 (not at all) to 3 (nearly every day). Higher scores indicate more severe anxiety.
Positive and Negative Affect Scale | Right before the first walking session, immediately after the sixth walking session, and one month after the sixth walking session.
  Positive and Negative Affect Scale measures positive and negative affect. The scale consists of 20 items, with 10 assessing positive affect (e.g., "passionate," "excited") and 10 assessing negative affect (e.g., "distressed," "upset"). Participants rated how strongly they experienced each emotion on a 5-point Likert scale, from 1 (very slightly or not at all) to 5 (very strongly).
Cognitive Flexibility Inventory | Right before the first walking session, immediately after the sixth walking session, and one month after the sixth walking session.
  Cognitive Flexibility Inventory measures individuals' ability to adapt to changing situations and consider multiple perspectives. Participants rated each item on a 5-point Likert scale, ranging from 1 (never) to 5 (always). Higher scores indicate greater cognitive flexibility.
Extended Inclusion of Nature in Self scale | Right before the first walking session, immediately after the sixth walking session, and one month after the sixth walking session.
  Extended Inclusion of Nature in Self scale measures individuals' perceived connection with nature, which refers to the degree to which individuals incorporate nature into their self-concept. Each item consists of seven pictures, scored on a 7-point scale, with higher scores indicating a stronger connection to nature.
Presence Scale | Immediately after each walking session.
  Presence Scale measures the state of being in which conditioned thinking ceases, and the mind is open, aware, non-reactive, and still; and often a witness of itself. Participants rated each item on a 7-point Likert scale, ranging from 1 (not at all) to 7 (completely). Higher scores indicate higher levels of Presence.

CONTACTS AND LOCATIONS:
Overall Officials: Xuanyi Wang, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Condon Hall, Seattle, Washington
  - Merrill Hall, Seattle, Washington